CLINICAL TRIAL: NCT05328661
Title: Pathophysiological Mechanisms of Trigeminal Neuralgia - Neurophysiological Assessment of the Blink-reflex
Acronym: TNBR
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Consultant in Neurology, Danish Headache Center
Other Study IDs: DanishHC180322Blink
Record Dates: First submitted 2022-03-18; First posted 2022-04-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Blinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blink reflex — The stimulator is directly connected to the right side of the frontal board. The sponge must be soaked in water or saline before being inserted into the stimulator. Dry them a bit to avoid leaking on the stimulator (it could create a bridge between the two poles). We want to stimulate the supraorbital nerve at its emergence from the eyebrow arch (the supraorbital foramen in the supra-orbital margin bone is easy to palpate 1 cm laterally to the root of the nose). We place the stimulator above the emergence of the supraorbital nerve, with the distal pole placed below. The final intensity of stimulation is generally between 5 to 10 mA, but higher intensities sometime are required.

SUMMARY:
This study aims to increase the understanding of the pathophysiology of trigeminal neuralgia by investigating the potential association between blink reflex abnormalities and phenotypical traits e.g. clinical characteristics and neuroimaging findings.

DETAILED DESCRIPTION:
We hypothesize:

Patients with classical trigeminal neuralgia have a prolonged latency and reduced amplitudes of the blink-reflex on the pain side compared to patients with idiopathic TN

The latency and amplitudes of the blink-reflex is normal in patients with idiopathic trigeminal neuralgia

Patients with concomitant persistent pain have a prolonged latency and reduced amplitudes of the blink reflex on the pain side compared to patients with pure paroxysmal TN

More men than women have a prolonged latency and reduced amplitudes of the blink reflex

Patients with neurovascular contact with morphological changes have prolonged latency and reduced amplitudes of the blink reflex compared to patients with simple neurovascular contact

Patients with secondary TN have prolonged latency and reduced amplitudes of the blink reflex compared to patients with simple neurovascular contact

Patients with neurovascular contact with morphological changes have prolonged latency and reduced amplitudes of the blink reflex on the pain side compared to the non-pain side

Study population

All patients with the diagnosis of primary or secondary trigeminal neuralgia, seen in the outpatient clinic at the Danish Headache Center will be screened for eligibility to participate the study. Clinical routine is not influenced by participation in this observational study. Patients will be offered the same treatment as patients not participating.

Setting

All patients with classic, idiopathic and symptomatic TN who have an appointment with a physician at the outpatient clinic at the Danish Headache Center as part of their work-up will, when they arrive at the center for their appointment, be asked if they want to participate in the study. The patients will be asked consecutively and there will be no prior recruitment of the patients. See recruitment below section 6.1. The study will not influence decisions regarding treatment of TN for the patients included in this protocol. Patients will be treated at the discretion of their own physician and the assessments listed below, are an integrated part of the clinical work-up and follow-up.

Assessments

Standardised data obtained from the medical chart

The following data will be obtained and registered from the medical chart of each patient that is included in the study:

Gender, date of birth, family history of TN or other facial pain

Duration and localization of TN, use of and response to previous medical treatments

Severity of pain at the time of examination - using Verbal Numerical Rating Scale (VNRS)

Location and trigger factors for TN

Previous neurosurgical treatment for TN

Additional concomitant diseases and medication

Type and dosage of TN related medication, if any

The result of the neurological exam.

Short interview on the examination day

On the day of the blink reflex examination, each patient will be asked by a trained biomedical laboratory scientist, nurse or medical student about the following:

Then the number of paroxysms

The current level of pain (VNRS)

The current dosage of TN medicine, will be on the day of neurophysiological assessments.

The trained personnel will not ask about the side of pain and will not know the result of the MRI evaluation, so they are blinded in terms of side of pain and what type of TN patient they investigate.

Neuroradiological assessment

The 3.0 Tesla MRI, performed according to a special TN protocol will be evaluated by a neuroradiologist, blinded for pain side. The neuro imaging data will be taken from the patient electronic journal. The following data will be registered:

Degree (no contact, simple contact, displacement/compression or atrophy of the nerve), location and type (arterial, venous or mixed) of NVC

Neurophysiological assessment (blink-reflex)

Electromyographic Recording:

We want to record signals from both eyes (see image). Channel 1: left eye. Channel 2: right eye

After connecting the cables to Channels 1 and 2 we can connect the electrodes to the black and red terminal wires: Black cable à active electrode: placed on the midline of the lower eyelid (orbicularis oculi muscles). Red cable à reference electrode: lateral to the eye (where the bone is superficial) We need one Green cable àground electrode: forehead or shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes with trigeminal neuralgia must meet the following inclusion criteria to be eligible for participation:

Age 18 years or older

Must be able to give Signed Informed Consent prior to study entry. Appendix X

Must fulfill the ICHD-3 diagnostic criteria1 for classical, idiopathic or secondary TN.

Has had a 3.0 Tesla MRI according to the trigeminal neuralgia protocol, maximum 2 years before or after the assessment of the blink-reflex.

Has had a semi-structured interview and neurological examination by the independent assessors, maximum 2 years before or after the assessment of the blink-reflex.

Exclusion Criteria:

* Subjects will be excluded if one of the following exclusion criteria is met:

If the patient is not able to give informed consent due to mental challenges

Previous neurosurgical treatment (microvascular decompression and/or ablative procedures) for trigeminal neuralgia

Bilateral trigeminal neuralgia

Symptomatic trigeminal neuralgia

Findings of sensory abnormalities detected at clinical neurological examination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Trigemnal neuralgia patients either with classic or idopathic TN
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Latency and amplitude of blink reflex on the pain side of classical trigeminal neuralgia patients. | 1 year
  We place the stimulator above the emergence of the supraorbital nerve, with the distal pole placed below. The subject could be in a sitting or supine position. He keeps his eyes opened and relaxed. The final intensity of stimulation is generally between 5to 10mA, but higher intensities sometime are required. We don't start from this intensity, but we increase it gradually from 2mA, in steps of 1-2mA. The time between consecutive stimuli must not be under 45 seconds, in order to avoid habituation. Before the stimuli is delivered, we look at the real-time activity box to be sure that the subject is relaxed. We aim to record at least 2-3 consecutive sweeps with a stable latency of the R1 and R2 components.

SECONDARY OUTCOMES:
Latency and amplitude of blink reflex on the pain side of idiopathic trigeminal neuralgia patients | 1 year
  We place the stimulator above the emergence of the supraorbital nerve, with the distal pole placed below. The subject could be in a sitting or supine position. He keeps his eyes opened and relaxed. The final intensity of stimulation is generally between 5to 10mA, but higher intensities sometime are required. We don't start from this intensity, but we increase it gradually from 2mA, in steps of 1-2mA. The time between consecutive stimuli must not be under 45 seconds, in order to avoid habituation. Before the stimuli is delivered, we look at the real-time activity box to be sure that the subject is relaxed. We aim to record at least 2-3 consecutive sweeps with a stable latency of the R1 and R2 components.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjerring B, Maarbjerg S, Heinskou T, Bendtsen L, Nikolic M, Grillo V, Icco R, Schytz HW. Comparison of the blink reflex in classical and idiopathic trigeminal neuralgia. Cephalalgia. 2023 Jul;43(7):3331024231191136. doi: 10.1177/03331024231191136. PMID 37525973